CLINICAL TRIAL: NCT01095679
Title: Assessment of the Effect of the GABA-B Receptor Agonist, Baclofen, on Hypoxia-induced Periodic Ventilation, in Healthy Subjects
Brief Title: Baclofen and Hypoxia-induced Periodic Ventilation
Acronym: PERIODIBAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P090207
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2009-12

CONDITIONS: CHEYNE Stokes Respiration
Keywords: CHEYNE Stokes respiration; Periodic ventilation; baclofen; hypoxia; healthy subject
MeSH Terms: conditions — Cheyne-Stokes Respiration; Hypoxia | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baclofen (Experimental)
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Breaking tablets of 10 mg of baclofen. Dosage and frequency : 5 mg 3 times a day for 3 days, then 10 mg 3 times a day for 3 days, then 15 mg 3 times a day for 3 days, then 20 mg 3 times a day for 3-5 days, then 15 mg 3 times a day for 1 day, then 10 mg 3 times a day for one day, then 5 mg 3 times a day for one day.
  Arms: Baclofen
Drug: Placebo — Breaking tablets of 10 mg of placebo. Dosage and frequency : 5 mg 3 times a day for 3 days, then 10 mg 3 times a day for 3 days, then 15 mg 3 times a day for 3 days, then 20 mg 3 times a day for 3-5 days, then 15 mg 3 times a day for 1 day, then 10 mg 3 times a day for one day, then 5 mg 3 times a day for one day.
  Arms: Placebo

SUMMARY:
Periodic ventilation that includes CHEYNE Stokes ventilation is a pathological pattern characterized by alternating periods of hyperpneas and apnea-hypopneas. It occurs generally during sleep, at high altitude and in hypoxic conditions in healthy subjects, and in some diseases like congestive heart failure. One study conducted on an animal model suggested that baclofen, a drug already used against spasticity in humans, could also be effective against periodic ventilation. The goal of the study is therefore to assess this hypothesis on hypoxia-induced periodic ventilation in healthy subjects during sleep.

DETAILED DESCRIPTION:
Rationale of the study:

Periodic ventilation, often called CHEYNE Stokes ventilation, results from a dysfunction of the mechanisms of the control of breathing. In this type of ventilation, alternating periods of hyperventilation and apneas and/or hypoventilation replace the normal regular pattern of breathing. Periodic ventilation occurs preferentially during sleep. It is responsible for decreases in arterial saturation in oxygen and for sleep fragmentation. There is currently no consensual treatment but non-invasive nocturnal mechanical ventilation is often used to bring the ventilatory pattern back to normal.

Periodic ventilation occurs in various conditions, the most frequent being cardiac failure. It also occurs in healthy subjects exposed to hypoxia or at high altitude.

The pathophysiology of periodic breathing remains poorly understood. Our hypothesis regarding the mechanisms of this abnormal ventilatory pattern is based on comparative physiology. Periodic ventilation is indeed the usual ventilatory pattern of many lower vertebrates. Moreover, even isolated in VITRO, the tadpole brainstem still produces a periodic ventilatory rhythm, characterized by clusters of ventilatory discharges. In this model, the agonist of the GABA-B receptor, the baclofen, transforms the periodic pattern into a regular one. Of note, the baclofen is already used in the treatment of some human diseases, especially against spasticity.

The hypothesis of the research project assumes that periodic ventilation in humans results from a neural reconfiguration of the networks that command breathing, leading them to produce an ancestral behavior. It also assumes that the baclofen woul reverse this phenomenon as it does in the model of the tadpole isolated brainstem.

The goal of the project is therefore to assess the effect of baclofen on hypoxia-induced periodic ventilation in healthy subjects during sleep. This is thus a pathophysiological study that aimed at demonstrating a concept before a possible clinical trial.

This study is pathophysiological study, conducted in healthy volunteers only.

Methods:

The subjects will sleep in hypoxic conditions, with a level of hypoxia similar to the one that is found at an altitude of 4000-4500 meters. A this altitude, the partial pressure of oxygen is approximately 90-100 mmHg. The hypoxic atmosphere will be created in a tent with an hypoxic generator (EVEREST Summit Hypoxic Generator, Hypoxic Systems, New York, NY, USA).

The electroencephalographic and electrocardiographic signals and the movements of the chest and of the abdomen will be recorded with a portable polysomnograph. The electromyogram of the chin and the ELECTRO Oculogram will also be recorded. These signals will permit to identify the sleep stages. The subjects will ware a face mask connected to a pneumotachometer for the recording of the ventilatory flow. Gas will also be sampled to measure the end tidal partial pressure of CO2.

Protocol:

Healthy volunteers will be enrolled after they will have given written informed consent. The subjects will be asked about their medical history and physical examination will be performed. Chest X-ray, electrocardiogram and pulmonary function tests will also be performed.

The subject will be asked not to sleep the night before each recording in hypoxic conditions (the hypoxic sessions). The recordings will be performed either during a nap in the afternoon or at night.

A first hypoxic session will be performed to identify the subjects who will develop periodic ventilation. Only those who will exhibit periodic ventilation during sleep will continue the study. They will be prescribed either baclofen or placebo (double blind, randomized). The posology will be progressively increased (over approximately 10 days) to reach 20 mg 3 times a day, during 3 to 5 days. A second hypoxic session will be performed under this treatment. Then the posology will be decreased over 3 days and a complete weaning will be performed during 5 to 10 days. The same protocol will be repeated, either with baclofen or placebo (depending of the previous run) and a third hypoxic session will be performed. The posology will then be decreased over 3 days and the study will be considered ended for the subject after 2 more days of complete weaning.

The maximum duration of the study for one subject will be 63 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Male
* Body mass index between 20 and 30 kg/m2
* Healthy (no known disease)
* No regular treatment except first grade antalgic drugs (e. g. ACETAMINOFEN)
* Written consent to participate in the study
* Health insurance

Exclusion Criteria:

* Intolerance to baclofen
* Tobacco, alcohol or drug consumption
* Past history of possible acute mountain sickness
* Regular treatment for any disease
* Claustrophobia
* Coronary disease
* Hypertension
* Cardiac failure
* Cardiac rhythm abnormalities
* Pulmonary hypertension
* Any pulmonary artery abnormality
* Any cardiac disease
* Past history of cerebral ischemia
* Past history of psychiatric disorder
* Any respiratory disease (including asthma)
* Leg arteriopathy
* Sickle cell anemia
* Renal insufficiency
* Migraine
* Diabetes
* Obesity
* Thalassemia
* Scoliosis
* Past history of phlebitis

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Decrease in the coefficient of variation of the period of the ventilatory cycle | During the second and the third session in hypoxia
  The primary outcome will be the decrease in the coefficient of variation of the period of the ventilatory cycle. The measures will be taken during the second and the third session in hypoxia. This means, for each subject, after having taken either placebo or 60 mg per day of Baclofen for 3-5 days.

SECONDARY OUTCOMES:
Decrease in the coefficient of variation of the tidal volume | During the second and the third session in hypoxia
  Decrease in the coefficient of variation of the tidal volume. The measures will be taken during the second and the third session in hypoxia. This means, for each subject, after having taken either placebo or 60 mg per day of Baclofen for 3-5 days.
Decrease in the coefficient of variation of the end tidal CO2 pressure | During the second and the third session in hypoxia
  Decrease in the coefficient of variation of the end tidal CO2 pressure. The measures will be taken during the second and the third session in hypoxia. This means, for each subject, after having taken either placebo or 60 mg per day of Baclofen for 3-5 days.
Decrease in the number of frequency compounds of the ventilatory flow | During the second and the third session in hypoxia
  Decrease in the number of frequency compounds of the ventilatory flow. The measures will be taken during the second and the third session in hypoxia. This means, for each subject, after having taken either placebo or 60 mg per day of Baclofen for 3-5 days.
Decrease in the apnea-hypopnea index | During the second and the third session in hypoxia
  Decrease in the apnea-hypopnea index. The measures will be taken during the second and the third session in hypoxia. This means, for each subject, after having taken either placebo or 60 mg per day of Baclofen for 3-5 days.
Decrease in the sleep fragmentation index | During the second and the third session in hypoxia
  Decrease in the sleep fragmentation index. The measures will be taken during the second and the third session in hypoxia. This means, for each subject, after having taken either placebo or 60 mg per day of Baclofen for 3-5 days.
Change in the non-linea dynamics of the ventilatory flow | During the second and the third session in hypoxia
  Change in the non-linea dynamics of the ventilatory flow. The measures will be taken during the second and the third session in hypoxia. This means, for each subject, after having taken either placebo or 60 mg per day of Baclofen for 3-5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Straus, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France